CLINICAL TRIAL: NCT04825626
Title: An Expanded Access IND to Evaluate the Safety and Preliminary Efficacy of Autologous HB-adMSCs for the Treatment of a Single Patient With Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Brief Title: An Expanded Access IND for the Treatment of Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Status: No longer available | Type: Expanded Access
Sponsor: Hope Biosciences Research Foundation (Industry)
Responsible Party: Sponsor
Other Study IDs: HBCIDP01
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: HB-adMSCs — Hope Biosciences adipose derived Mesenchymal Stem Cells.
  Other Names: MSCs

SUMMARY:
This is an Individual Patient Expanded Access IND to evaluate the safety and preliminary efficacy of autologous HB-adMSCs for treating a single patient Chronic Inflammatory Demyelinating Polyneuropathy, CIDP. The expanded access program will include a screening period of up to 28 days, a 44-week treatment period, a safety follow-up at 50, and a 52-week end-of-study visit.

DETAILED DESCRIPTION:
An informed consent form will be given to the participant, who will sign before any procedures.

The informed consent form will include information about this expanded access and all the aspects considered during this process. The participant is required to complete the subsequent visits after they have given their informed consent.

* Visit 1 - Screening during this period, the principal investigator will determine whether the screened participant is eligible and whether the next visit can be scheduled. Once the principal investigator has evaluated the eligibility (up to 28 days), the patient will be scheduled for the first infusion.
* Visit 2 - Infusion 1 (Baseline): this visit will be a starting point for comparing participant's data. During this visit, the patient will receive the 1st investigational product via intravenous infusion, with rigorous monitoring of vital signs for a total of 2 hours.
* Visit 3 to 12 - During these visits, the patient will receive intravenous infusions of HB- adMSCs while her vital signs are precisely monitored for a total of 2 hours.
* Follow-Up Phone Call - During this safety follow-up phone call, the principal investigator will evaluate the safety of the investigational product by conducting several assessments described in the Schedule of Assessments table.
* End of Study - At the end of the expanded access program visit, the principal investigator will conduct various evaluations to determine the patient's physical condition and assess whether there have been any safety events resulting from the participation in the expanded access program.

ELIGIBILITY:
* Inclusion Criteria

  * Patient diagnosed with Chronic Inflammatory Demyelinating Polyneuropathy, CIDP, with documented medical records.
  * Patient must have banked his stem cells at Hope Biosciences LLC.
* Exclusion Criteria

  * The patient has any active infection requiring medications.
  * The patient has any suicidal ideation during the screening visit or at any point during the study.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Djamchid Lotfi, MD, Principal Investigator — Hope Biosciences Stem Cell Research Foundation
Locations (1):
- Hope Biosciences Stem Cell Research Foundation, Sugar Land, Texas, United States